CLINICAL TRIAL: NCT00644852
Title: Medical Chart Review of Patients on Long-term Treatment With Long-acting Injectable Risperidone
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CR013993
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective disorder; Risperidone long-acting injectable, Long-term evaluation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- 001
  Interventions: Other: Retrospective chart review study

INTERVENTIONS:
Other: Retrospective chart review study — Retrospective study chart review long acting risperidone

SUMMARY:
The purpose of the study is to evaluate the characteristics, clinical responses, and safety issues of patients receiving long-term treatment of Risperidone long-acting injectable. The goal is to evaluate patient outcomes based on pre-existing risk or disease factors and past medication use.

DETAILED DESCRIPTION:
This is an Observational, retrospective study on the use of Risperidone long-acting injectable. The purpose of the study is to evaluate the characteristics, clinical responses, and safety issues of patients receiving long-term treatment of Risperidone. Patient outcomes will be evaluated based on pre-existing risk or disease factors and past medication use. Data will be collected from medical charts and other available medical records from one year prior to risperidone treatment until discontinuation of risperidone long acting injectable. The study will compare the number of days hospitalized for reasons relating to psychosis before and after treatment with risperidone long-acting injectable. Information about past use of anti-psychotic medications will be collected. The occurrence and frequency of adverse events [Extra-Pyramidal Symptoms (EPS) - the abnormal body movements sometimes associated with antipsychotic medications, body weight changes, drowsiness, sexual problems] and the dose or change in dose of Risperidone long-acting injectable will also be collected. The study will also investigate the relapse rate and the hospitalization rate before and after treatment. It is a chart review type of study. No study drug has been used in the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia or Schizoaffective disorder by DSM-IV-TR criteria
* Patients who used to be treated with Risperidone long-acting injectable regularly for at least 3 months
* Patients whose medical charts or other medical records are available

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll patients with diagnosis of Schizophrenia or Schizoaffective disorder by DSM-IV-TR criteria and who have ever been treated with risperidone long-acting injectable for more than 3 months.
Sampling Method: Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2007-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Compare the number of days hospitalized for reasons relating to psychosis before and after treatment with risperidone long-acting injectable. | From one year prior to risperidone treatment until discontinuation of risperidone long acting injectable.

SECONDARY OUTCOMES:
Compare the Relapse Rate and the Hospitalization Rate before patients were treated with risperidone long-acting injectable | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan, Ltd. Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd